CLINICAL TRIAL: NCT03680313
Title: Cardio-ankle Vascular Index (CAVI) in Hypertension Patients After One Year of Treatment
Status: Completed | Type: Observational
Sponsor: Hanoi Medical University (Other)
Responsible Party: Principal Investigator, Bui My Hanh, Director, Science Research and International Cooperation Unit, Hanoi Medical University
Other Study IDs: HMU16225
Record Dates: First submitted 2018-09-18; First posted 2018-09-21 (Actual); Last update posted 2018-09-21 (Actual); Status verified 2018-09

CONDITIONS: Hypertension
Keywords: Cardio-ankle vascular index (CAVI)
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hypertension group: All adult patients (above 18 year of age) were recruited between May, 2016 and June 2017, at Duc Giang General Hospital. The inclusion criteria are as followed:
  * Patients have never been diagnosed with hypertension.
  * Has been diagnosed with primary hypertension, but not take any treatment.
  Interventions: Procedure: Hypertension outpatient treatment
- Control group: A group of normal people with the similar age to hypertension group was recruited as control group at the same time

INTERVENTIONS:
Procedure: Hypertension outpatient treatment — Patients who have been diagnosed with primary hypertension and meet the conditions of the study will receive outpatient treatment
  Groups: Hypertension group

SUMMARY:
This study aimed to evaluate the role of the cardio-ankle vascular index (CAVI) in evaluating arterial stiffness changes, the degree of atherosclerosis in patients with hypertension after 1 year of treatment and analysis the correlation between CAVI and cardiovascular risk factors.

ELIGIBILITY:
Inclusion Criteria:

* Patients have never been diagnosed with hypertension.
* Patients have been diagnosed with primary hypertension, but not take any treatment

Exclusion Criteria:

* Cases with non-primary hypertension or suffering from cardiovascular complications such as myocardial infarction, cerebral stroke, vascular disease, severe heart failure (EF<1) in the time of measurement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The eligible patients were prospectively monitored to evaluate CAVI in hypertension treatment for every 3 months. All participants will be asked directly medical history, clinical examination and performed blood pressure measurement thoroughly. All clinical information will be retained in medical record.
Sampling Method: Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-06-01 (Actual)

PRIMARY OUTCOMES:
CAVI score in hypertension group after one year of treatment | 1 year
  CAVI score of patients who achieved their target blood pressure after one year of hypertension treatment

SECONDARY OUTCOMES:
Correlation between CAVI and smoking status | 1 year
  Evaluating correlation between CAVI score and smoking status in hypertension patients
Correlation between CAVI and overweight status | 1 year
  Evaluating correlation between CAVI score and overweight status in hypertension patients
Correlation between CAVI and diabetes status | 1 year
  Evaluating correlation between CAVI score and diabetes status in hypertension patients
Correlation between CAVI and dislypidemia status | 1 year
  Evaluating correlation between CAVI score and dyslipidemia status in hypertension patients

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code